CLINICAL TRIAL: NCT04884568
Title: An Open, Non-comparative, Post-market Clinical Follow-up Investigation to Confirm Performance and Safety of Exufiber When Used as Intended on Donor Sites
Brief Title: Confirm Performance and Safety of Exufiber When Used as Intended on Donor Sites
Acronym: ExuDS01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ExuDS01
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Acute Wound; Donor Site; Split Skin Graft
Keywords: Post Market Clinical Follow-up; Exufiber; Gelling fibre dressing

STUDY DESIGN:
Intervention Model Description: Single group of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exufiber (Experimental): This is an open, non-randomised , single arm study
  Interventions: Device: Exufiber

INTERVENTIONS:
Device: Exufiber — Wound dressed with Exufiber for up to 21 days.

SUMMARY:
This is a single-centre prospective, open, non-comparative, Post-Market Clinical Follow-up (PMCF) investigation to confirm performance and safety of Exufiber® (Gelling fibre dressing) when used as intended on donor sites through assessment of wound progression from baseline to the subject´s last visit.

DETAILED DESCRIPTION:
A single-centre prospective, open, non-comparative, PMCF investigation to confirm performance and safety of Exufiber® (gelling fibre dressing) when used as intended on donor sites. The investigation will include eligible subjects undergoing split skin graft transplantation for harvesting of a partial-thickness skin graft, i.e. excision of the epidermis and part of the dermis. After the study inclusion (baseline) the patient will go through the split skin graft transplantation following application of the Exufiber® dressing, Mepilex®(non-border) dressing, and any third dressing as required on the donor site. Each subject will thereafter be followed up on days 3, 14, and 21 prior completion in the study.

A subject may complete the study prior to or on day 14 as well as in between day 14 and day 21 if the donor site is healed. Wound healing progression will be determined by the investigator/designee and assessed as:

* 100% re-epithelialisation including small residual scabs/blisters and open areas less than 1 cm within an otherwise fully re-epithelialised area, and/or
* less than 100% re-epithelialization but to the extent that the Exufiber dressing is not required anymore

If the donor site is not healed and the donor site is dry and therefor not treatable with Exufiber the patient will be treated according to clinical praxis and followed for outcomes on the following visits.

Approximately 34 eligible subjects will be included in one centre in Sweden.

The primary performance endpoint will be progression of donor site wound from baseline to last visit when Exufiber is used, up to 21 days.

Wound progression will be determined by the investigator/designee and will be assessed as one of the following three outcomes:

* Deteriorated
* No change
* Improved

ELIGIBILITY:
Inclusion Criteria:

1. Female or male ≥18 years old.
2. Scheduled for a split skin graft transplantation of a partial thickness graft at a healthy and intact location at the thigh.
3. Planned hospitalization for at least 3 days post-transplantation.
4. Size of donor site treatable with an 15cm x 15cm Exufiber, with 2-3 cm additional overlap to dry surrounding skin.
5. Provision of written informed consent

Exclusion Criteria:

1. Burn injury of ≥20% of total body surface area.
2. Diagnosed with paraplegia.
3. Harvested graft from the same donor site location before.
4. Donor sites not to be harvested with dermatome
5. Pregnancy or lactation at the time of screening.
6. Known allergy/hypersensitivity to Exufiber, Mepilex or other components/products used in this investigation.
7. Participating in other ongoing clinical investigation that may impact the outcome of this investigation based on the judgement of the investigator.
8. Not able to read or understand Swedish.
9. Any other conditions that according to the investigator may make follow-up or investigation inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Change in wound progress | Day 14(-1 day), Day 21(+-1 day)
  Wound progress compared between each visit up to final visit and assessed as:
  * Deteriorated
  * No change
  * Improved

SECONDARY OUTCOMES:
Change in wound progress | Day 14(-1 day)
  Wound progress compared between baseline and final visit up to 14 days and assessed as:
  * Deteriorated
  * No change
  * Improved
Wound healing progress | Day 14(-1 day), Day 21(+-1 day)
  Wound healing progress will be assessed between baseline and final visit and assesed as:
  - Rating percentage (%) re-epithelialisation using a visual score (0-100%). 0% is equal to no re-epithelialisation and 100% is equal to fully re-epithelialised.
Follow-up assessment of wound healing when treated according to clinical praxis | Day 21(+-1 day)
  Wound healing progress for subjects treated according to clinical praxis when wound is not healed and not treatable with Exufiber (dry wound) will be followed up at the final visit and assessed as:
  - Rating percentage (%) re-epithelialisation using a visual score (0-100%). 0% is equal to no re-epithelialisation and 100% is equal to fully re-epithelialised.
Wound size | Day 14(-1 day)
  Wound dimension/size assessed as area using following assessments:
  Width (mm) Length (mm)
Change in exudate amount and type | Day 14(-1 day), Day 21(+- 1 day)
  Evaluation of the amount of wound exudate and the exudate type at each follow-up visit using the variables below:
  Exudate amount:
  * High
  * Moderate
  * Low
  * None
  Exudate type:
  * Serous
  * Serousanguinous
  * Sanguinous
  * Purulent
  * N/A
Local infection | Day 14(-1 day), Day 21(+- 1 day)
  Presence of signs of local wound infection determined at each follow-up visit, using the variables listed below:
  * Swelling
  * Redness
  * Heat
  * Fever
  * Pain
  * Foul odour
Subject's pain | Day 14(-1 day), Day 21(+- 1 day)
  Subject's pain captured using a numeric rating scale(NRS) at each follow-up visit where the patient verbally grade his/her pain on a level from 0 to 10, where 0 indicates no pain and 10 the worst imaginable pain for the subject. The NRS will be used at the following occasions:
  * Pain before dressing removal
  * Pain when removing Mepilex (secondary dressing)
  * Pain when removing Exufiber
Subject's itching | Day 14(-1 day), Day 21(+- 1 day)
  Subject's itching captured at each follow-up visit using the NRS scale where the patient verbally grade their itching on a level from 0 to 10, where 0 indicates no itching and 10 the worst imaginable itching for the subject.
  The subject will answer the NRS question, about itching intensity, just before dressing removal.
Ability of dressing to absorb blood | Day 21(+-1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing and their ability to absorb blood using the variables below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ability of dressing to absorb exudate | Day 21(+-1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing and their ability to absorb exudate using the variables below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ability of dressing to retain exudate | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to asses performance of the primary and secondary dressing and its ability to retain exudate using the variables below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ability of the dressing to retain blood | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing and their ability to retain blood using the variables below:
  Very poor
  Poor
  Good
  Very good
  N/A
Exudate leakage | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing in regards to exudate leakage, using the variables below:
  Major
  Minor
  None
  N/A
Blood leakage | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing in regards to blood leakage, using the variables below:
  Major
  Minor
  None
  N/A
Ability of dressing to stay in place | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary and secondary dressing and their ability to stay in place, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ease of handling | Day 21(+-1 day)
  A subjective measurement captured at the final visit to assess the handling of the primary dressing and ease of dressing application, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ease of dressing removal | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess the ease of removal of the primary dressing, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing conformability | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary dressing and its ability to conform, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing integrity | Day 21(+- 1 day)
  A subjective measurement captured at the final visit to assess performance of the primary dressing and its ability to maintain integrity by being removed in one piece, using the variables below:
  Very poor
  Poor
  Good
  Very good
  N/A
Comfort and experience | Day 21(+-1 day)
  The subject's perception of comfort and experience of the primary dressing will be captured at the final visit by asking questions to the subject :
  * Comfort during wear of the dressing
    * Very Poor
    * Poor
    * Good
    * Very Good
    * N/A
  * Experience during dressing change
    * Very Poor
    * Poor
    * Good
    * Very Good
    * N/A
  * Overall impression of the dressing
    * Very Poor
    * Poor
    * Good
    * Very Good
    * N/A
Subject's quality of life assessment | Day 21(+- 1 day)
  Impact of everyday life will be captured at the final visit through a NRS scale where the subject will grade how much the treatment has affected the his/her daily life. 0 is equal to no influence and 10 to considerable influence on everyday life or unbearable.
  If replying >0, the subject will state the presence or absence of the following causes:
  * Leakage of dressing
  * Impaired mobility
  * Difficulties in getting dressed
  * Pain
  * Odor
Dressing wear time | Day 3, Day 14(-1 day), Day 21(+- 1 day)
  Dressing wear time of the primary and secondary dressings will be captured in a Dressing log from baseline until final visit including unscheduled extra visits.
pH level measurement | Day 3
  Levels of pH in the wound bed will be captured if it is deemed necessary to change both primary and secondary dressings, using pH indicator paper sticks.

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University Hospital /Department of Hand and Plastic Surgery & Burn Center, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No